CLINICAL TRIAL: NCT02717065
Title: Variability of Tinnitus Characterization Tools and Investigation of Audiovisual Integration in Tinnitus Perception
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Personnel and funding was no longer available
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1512M81434
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Tinnitus
Keywords: Neuromodulation; Noninvasive; Plasticity; Hearing; Hyperacusis
MeSH Terms: conditions — Tinnitus; Hyperacusis | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Characterization, Audiovisual (Experimental): Characterization: Tinnitus characterization tools (Minimal Masking Level, Tinnitus Functional Index, Tinnitus Handicap Inventory, and Subjective rating scale) are assessed in an individual over time to determine baseline variability.
  Audiovisual: The individual will watch a series of silent videos of a person speaking, both with and without a tone matched to their tinnitus as well as videos of a still face with and without the matched tone.
  Interventions: Other: Tone; Other: Video

INTERVENTIONS:
Other: Tone — Band-limited white noise stimulus or frequency-matched tone presented at a comfortable loudness level via headphones or earphones.
Other: Video — Silent video recording of a person speaking or a still face with an expanding circle over the mouth presented on a computer or tablet screen.

SUMMARY:
Characterizing the nature and severity of tinnitus in individuals presents a particular challenge. The nature of the sound (loudness and pitch) is not necessarily indicative of the effect on quality of life. Different methods are used to measure each parameter. Loudness is measured using a technique called "minimum masking," in which the subject is presented with a broadband white noise and asked to adjust the loudness level until they can no longer hear their tinnitus. Severity of tinnitus is commonly characterized using two questionnaires: the Tinnitus Handicap Inventory (THI) and the Tinnitus Functional Index (TFI). These questionnaires assess the perceived severity of the tinnitus and the effect on everyday activities and quality of life. A visual analog scale (a scale from 0-10) is used as a general subjective measurement of tinnitus severity. In the first part of this study, we will measure each of these parameters over a series of sessions to establish a baseline variability for each individual.

The second part will look at the influence of context-specific visual information on auditory perception. This involves watching silent videos of a person speaking, with and without an additional tone designed to match the subject's tinnitus. The effect of this audiovisual feedback on the subject's perception of tinnitus will be assessed using a subjective rating scale and the minimum masking task.

DETAILED DESCRIPTION:
This study is not specifically seeking to treat tinnitus, but is designed to investigate various parameters that can alter the tinnitus percept. Findings from this study will help identify parameters that can be more effective at decreasing or fully suppressing the tinnitus percept that will be systematically explored in a follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Have subjective, non-pulsatile and bothersome tinnitus
* Ability to give informed consent and understand study objectives and procedures in English
* Willing and able to understand and comply with all study-related procedures
* Will not start any new tinnitus treatment during the study

Exclusion Criteria:

* Substantial hearing loss or hyperacusis that may interfere with the study
* Medical history of other ear or brain disorders
* Pregnant or currently breast-feeding (we need to give all female subjects a pregnancy test because pregnant females and unborn children require extra protection for their safety)
* Any handicap that prevents the subject from reliably performing the tests, such as blindness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Change in Minimal Masking Level | Change in baseline level at an expected average of 1 minute and 1.5 hours after testing paradigm.
  A narrowband noise (from 2-12 kHz) is presented to the tinnitus ear and the minimum sound level (in decibel sound pressure level, decibel SPL) is determined that completely masks the tinnitus percept.
Change in Tinnitus Rating (0-10, 10 being worst) | Change in baseline rating at an expected average of 4 minutes and 1.5 hours after testing paradigm
  the subject rates the disturbance or bothering nature of the tinnitus.

SECONDARY OUTCOMES:
Change in Tinnitus Functional Index Questionnaire Score | Change from baseline score at an expected average of 5 minutes and 1.5 hours after testing paradigm
  A series of questions to assess the quality and bothering nature of the tinnitus, which is then quantified into a single score.
Change in Tinnitus Handicap Inventory Questionnaire Score | Change from baseline score at an expected average of 5 minutes and 1.5 hours after testing paradigm
  A series of questions to assess the quality and bothering nature of the tinnitus, which is then quantified into a single score.
Change in Tinnitus Subjective Description | Change in baseline description at an expected average of 5 minutes and 1.5 hours after testing paradigm
  The subject describes the quality, characteristics, and bothering nature of the tinnitus.

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Lim, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Nils Hasselmo Hall, 6-105, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No